CLINICAL TRIAL: NCT05855837
Title: Appetite Responses to Cereal Products: A Randomized Controlled Trial
Brief Title: Appetite Responses to Cereal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/03/21
Record Dates: First submitted 2023-05-02; First posted 2023-05-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: Satisfaction, Consumer
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cereal Product 1 (Experimental): Ready to Eat Cereal Product 1 with 6 oz of skim milk
  Interventions: Other: Ready to Eat Cereal
- Cereal Product 2 (Experimental): Ready to Eat Cereal Product 2 with 6 oz of skim milk
  Interventions: Other: Ready to Eat Cereal
- Control (No Intervention): No intervention (i.e., no food provided)

INTERVENTIONS:
Other: Ready to Eat Cereal — Cereal products available in retail stores
  Arms: Cereal Product 1; Cereal Product 2

SUMMARY:
The purpose of this clinical trial is to investigate appetite responses to 2 cereal products in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-70 years old
* Habitual cereal consumers (at least several times per month)
* Body mass index 18.5-24.9 kg/m2 (based on self-reported weight and height
* Understand and willing to follow the study procedures
* Willing to drink skim milk
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the study
* Willing to abstain from strenuous exercise and consuming alcoholic drinks 24 hours before the test day
* Willing to provide Informed Consent to participate in the study

Exclusion Criteria:

* Pregnant or lactating women, or women who are planning to become pregnant during the study
* Known food allergies, sensitivities, or intolerance to any food or food ingredients
* Participation in another clinical trial for food, investigational drug, nutritional supplement, or lifestyle modification
* Taking medication(s) that affect appetite, metabolism or blood pressure
* Presence of acute diseases or infection
* Presence or history of chronic diseases
* Diagnosed with an eating disorder
* Restraint eaters as determined by score >4 from the Dutch Eating Behavior Questionnaire
* Lost or gained 5 or more pounds in the past 3 months
* On a weight loss diet or undergoing intermittent fasting
* COVID-19 infection within the past 3 months
* Subjects who do not eat cereal products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Hunger 0-240 minutes | 240 minutes
  Visual Analogue Scale for "how hungry are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more hunger. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a lower mm change from baseline indicates a better outcome.
Visual Analogue Scale for Fullness 0-240 minutes | 240 min
  Visual Analogue Scale for "how full are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more fullness. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a higher mm change from baseline indicates a better outcome.
Visual Analogue Scale for Satiation 0-240 minutes | 0-240 min
  Visual Analogue Scale for "how satiated are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more satiation. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a higher mm change from baseline indicates a better outcome.
Visual Analogue Scale for Desire to Eat 0-240 minutes | 240 min
  Visual Analogue Scale for "how strong is your desire to eat right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more desire to eat. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a lower mm change from baseline indicates a better outcome.
Visual Analogue Scale for Prospective Consumption 0-240 minutes | 240 min
  Visual Analogue Scale for "how much do you think you can eat right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more prospective consumption. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a lower mm change from baseline indicates a better outcome.
Visual Analogue Scale for Satisfaction 0-240 minutes | 240 min
  Visual Analogue Scale for "how satisfied are you right now?" is scored from 0-100 millimeters (mm), whereby a higher mm indicates more satisfaction. Comparing change from 0 minutes (baseline) to 240 minutes, whereby a higher mm change from baseline indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Remote study, no physical facility, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No